CLINICAL TRIAL: NCT06345625
Title: Gait and Postural Balance Analysis During Head-motion Perturbed Standing and Walking in Older Adults - a Multisensory Approach by Use of Mixed-reality
Brief Title: Gait and Postural Balance Analysis During Head-motion Perturbed Standing and Walking in Older Adults
Acronym: BALANCAR
Status: Recruiting | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Ann Hallemans, Associate Professor, Universiteit Antwerpen
Other Study IDs: 6012
Record Dates: First submitted 2024-03-05; First posted 2024-04-03 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Aged; Accidental Fall; Postural Balance; Gait
Keywords: older adults; Sensorimotor integration; visual tracking while walking
MeSH Terms: interventions — Sensation; Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fallers: Community dwelling older adults with an age above 65 years. A participant is categorized as faller in case of a history of ≥2 falls in the previous 12 months and with identified high fall risk on the TUG (i.e., completion time ≥13.5 seconds). A fall is defined as an event that results in a person coming to rest inadvertently on the ground/floor/other lower level (WHO, 2021). Asyncopal fall, identified through the report of a loss of consciousness during the fall, has a different etiology and therefore will not be counted as a fall (Ang et al., 2020).
  Interventions: Diagnostic Test: Cognition; Diagnostic Test: Sensory function; Diagnostic Test: Frailty; Other: Biomechanical movement analysis; Other: Screening; Other: Follow up
- Non-Fallers: Community dwelling older adults with an age above 65 years. A participant is included as non-faller in case of a history of 0 falls in the previous 12 months and without an identified fall risk on the TUG test (i.e., completion time ≤13.5 seconds).
  Interventions: Diagnostic Test: Cognition; Diagnostic Test: Sensory function; Diagnostic Test: Frailty; Other: Biomechanical movement analysis; Other: Screening; Other: Follow up

INTERVENTIONS:
Diagnostic Test: Cognition — 1. The CatchU® app quantitatively and objectively measures the ability to integrate visual-somatosensory information using reaction time test data.
  2. Digit Symbol Substitution test assesses processing speed and attention by requiring individuals to match symbols with corresponding numbers within a specified time frame.
  3. Trail Making Test part 1 and 2: assesses cognitive flexibility, visual attention, and task-switching by having individuals connect numbered circles in sequence (part 1) and then alternate between numbers and letters (Part 2).
  4. Go/No Go test measures an individual's ability to inhibit a prepotent response (No-Go) and execute a response when required (Go). This test provides insights into executive functioning, particularly inhibitory control.
Diagnostic Test: Sensory function — 1. Cervical Sensorimotor control will be measured through a wireless wearable sensor 3D-cervical trainer by Sensamove on the placed on the head of the participant. The 3DCT registers cervical position sense by the Head Repositioning Accuracy test where the subject must relocate the head to the previously memorized (neutral) head position with the eyes closed and the joint position error degrees are registered. Cervical movement sense is examined using 'The Fly'-test where the subject ought to follow a movement pattern displayed on the screen in front of them. The movement of the neck-head unit is there upon tracked by the 3DCT and projected on the screen.
  2. Vestibular function will be assessed through 3D-video Head Impulse Testing (vHIT), examining the state of the three semicircular canals by delivering the vestibulo-ocular reflex (vor) gain and vor gain asymmetry.
  3. For the assessment of static and dynamic visual acuity, functional Head Impulse Testing (fHIT) will be used.
Diagnostic Test: Frailty — Frailty will be assessed using the Fried criteria, comprising 5 categories (each accounting for 1 point if scored positive): Unintentional weight loss (interview), weakness (grip strength with hand-held dynamometer), poor endurance and energy (two statements of the CES-D Depression Scale), slowness (walking speed over 15ft through gait analysis) and low physical activity level (Minnesota Leisure Time Activity questionnaire)(Fried et al., 2001).
Other: Biomechanical movement analysis — Markers will be placed on the predefined anatomical locations and surface electrodes for electromyography will be applied at the predefined muscle locations following the SENIAM-guidelines. The Microsoft HoloLens 2 is fixated on the participant's head which will, on one hand, provide the cue to the participant for the head movement and on the other hand track eye and head movements. A safety harness is attached to the body and the ceiling of the lab. At the start of the trial, the subject will see a projection by the HoloLens 2 on the real environment moving to the left; right; upward; downward (cue in randomized order) which the participant is ought to follow with eyes and head. First while standing still and second while walking the 10-meter overground walkway at a self-preferred walking speed.
Other: Screening — The researcher will visit the possible participants (at their home, community centre, etc.) and after written consent on screening procedure is provided, the tests for eligibility will be performed.
  1. Interview: asking about age (years), gender (male/female), medical history and the number of falls in the last 12 months .
  2. Timed Up-and-Go (TUG) to check walking ability. TUG is a sensitive and specific measure for identifying risk for falls (Shumway-Cook et al., 2000).
Other: Follow up — Participants are followed up for 12 months. They fill in a fall diary and telephone reminders will be performed monthly to encourage participants to complete and return their diaries.

SUMMARY:
The main aim of this study is to unravel the biomechanics of postural balance reactions during head-motion perturbed standing and walking in older adults who fall, while integrating the influence of frailty, sensory functioning and cognitive processing.

DETAILED DESCRIPTION:
Older adults above 65 years old experience falls at a rate of 20-40% annually, with women being more affected than men. Unintentional falls are the second leading cause of accidental injury death and a major contributor to disability levels worldwide. Falls pose an even bigger burden on society in the future due to the increasing number of older adults and the higher prevalence of falls as people age. Gait and balance instability are major risk and causative factors for falls in older adults. As people age, their stability decreases. This is evident in the careful way that older adults walk. To prevent and predict falls, it is essential to understand how humans maintain their stability during locomotor activities.

Balance disruptions are typically not caused by walking itself, but rather by internal or external disturbances or the performance of multiple tasks simultaneously. In daily life, people often face complex situations that require high levels of sensory input and cognitive processing. This can be especially challenging when also trying to maintain a safe walking pattern, such as when checking the environment before crossing the street. This task requires coordinated movement of both the head and eyes to track moving objects. Gaze control requires accurate cognitive processing, including multisensory integration, attention, executive functioning, and motor responses to coordinate eye and head movements.

Older adults use different strategies than younger adults to control head movement for stabilizing their head during walking. Therefore, changes in head position may affect gait stability differently in older adults. Ageing can cause frailty, decline in sensorimotor and cognitive abilities, and a reduced capacity to adjust gait to changing environments. These changes may increase the risk of falls in older adults. However, research on these issues is currently insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* an age of 65 years or above

Exclusion Criteria:

* age < 65 years
* medical history encompassing diagnosed vestibulopathy, orthostatic hypotension, peripheral neuropathy, limb amputation, neurological or neuromuscular disorders affecting balance, diagnosed neck disorders affecting sensorimotor control, blindness, deafness
* a full-time walking aid is indispensable.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community dwelling older adults with an age of 65 years or above
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Spatio-temporal parameters of gait | baseline
  step length and width (cm)
Foot placement estimator | baseline
  measure which estimates where the foot should be placed for stable gait
Onset latency | baseline
  latency in msec between onset of movements and activation recorded by surface EMG of bilateral m. Erector Spinae (trunk stabilization), m. Gluteus medius (hip strategy), m. Tibialis anterior and m. Soleus (ankle strategy)
Peak amplitude | baseline
  peak amplitude in microvolts of the surface EMG of bilateral m. Erector Spinae (trunk stabilization), m. Gluteus medius (hip strategy), m. Tibialis anterior and m. Soleus (ankle strategy)
Fixation duration | baseline
  Duration of fixation of the eyes on target, measured by the Hololens 2
Gain | baseline
  Accuracy of the fixation of the eyes on target as measured by the Hololens 2
Latency | baseline
  Latency in msec between the movement of the target and the movement of the eyes and the head when following the target as measured by the Hololens 2.
Fall characteristics | monthly during 12 months of follow-up
  Fall diaries provide information on occurrence and number of falls, activity preceding a fall, cause of fall, obtained injuries and potential care that was received.

SECONDARY OUTCOMES:
Multisensory integration | baseline
  reaction times in visual/sensory vs. visuo-sensory conditions (ratio, in %) measured with CatchU app
Digit symbol substitution test | baseline
  number of correct symbol-digit pairs completed
Trail making test | baseline
  Time to complete part A vs. B (ratio in seconds)
Go/No Go test | baseline
  Accuracy (number of correct responses)
Head Repositioning Accuracy | baseline
  joint position error in degrees
Fly test | baseline
  directional accuracy (in %) of movement
Fly test | baseline
  Amplitude (in mm) of movement
vHIT | baseline
  VOR-gain and VOR-gain asymmetry in %
fHIT | baseline
  statfHIT (Static visual acuity): logMAR-score and dynfHIT (Dynamic visual acuity): % correct responses
Frailty | baseline
  Fried criteria: Frailty level (categorical): non-frail (0/5), pre-frail( 1-2/5) or frail (≥3/5)

OTHER OUTCOMES:
Age | Screening before inclusion
  age in years
Gender | Screening before inclusion
  male, female or other
Medical history | Screening before inclusion
  presence or absence of diagnosed vestibulopathy, orthostatic hypotension, peripheral neuropathy, limb amputation, neurological/ or neuromuscular disorders affecting balance, neck disorders affecting sensorimotor control, blindness, deafness and if a full-time walking aid is indispensable
Fall history | Screening before inclusion
  number of falls in last 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Hallemans, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided